CLINICAL TRIAL: NCT00006138
Title: Diagnostic Pilot Study of Dual Energy Absorptiometry in the Detection of Osteopenia or Osteoporosis in Patients With Thalassemia Major
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Children's Hospital of Philadelphia (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/15314; CHP-IRB-1998-6-1502; CHP-GCRC-1655
Record Dates: First submitted 2000-08-03; First posted 2000-08-04 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-10

CONDITIONS: Osteoporosis; Thalassemia Major; Osteopenia
Keywords: disease-related problem/condition; genetic diseases and dysmorphic syndromes; hematologic disorders; osteoporosis; rare disease; thalassemia major
MeSH Terms: conditions — Osteoporosis; beta-Thalassemia; Bone Diseases, Metabolic; Genetic Diseases, Inborn; Hematologic Diseases; Rare Diseases

SUMMARY:
OBJECTIVES:

I. Determine the frequency and severity of osteopenia and osteoporosis in patients with thalassemia major who undergo dual energy x-ray absorptiometry, and correlate these findings with other relevant endocrinologic measurements.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients undergo dual energy x-ray absorptiometry for bone density measurements, height (sitting and standing) and weight measurements, comprehensive endocrinologic examination, and assessment of the severity of iron overload at baseline, and then at years 1 and 2.

ELIGIBILITY:
* Diagnosis of thalassemia major with iron overload
* Not pregnant
* Negative pregnancy test

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35
Dates: Start 1998-06; Study Completion 2000-08

CONTACTS AND LOCATIONS:
Overall Officials: Alan Richard Cohen, Study Chair — Children's Hospital of Philadelphia